CLINICAL TRIAL: NCT00893191
Title: The Effect of Sildenafil on Sleep-Disordered Breathing in Obese Patients With Sexual Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Isaac Shpirer, Asaf Harofeh Medical Center
Other Study IDs: 39/09
Record Dates: First submitted 2009-05-03; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Sildenafil; Sleep Apnea; Sexual Dysfunction; Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Sexual Dysfunction, Physiological; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Sildenafil: Treated with 50 mg of Sildenafil at night
- Placebo: Treated with placebo at night

SUMMARY:
Sildenafil has been shown to aggravate sleep-disordered breathing in patients with severe obstructive sleep apnea. The aim of the present study is to examine the frequency of sleep-disordered breathing in obese patients who are candidates for treatment with sildenafil for sexual dysfunction. In addition we wish to assess the effect of sildenafil on sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Age - 40-65 years
* BMI equal to or over 30

Exclusion Criteria:

* A known cardiorespiratory, liver or kidney disease
* Treatment with nitrates or alfa blockers
* Performed polysomnography in the past

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 healthy males aged 40 - 65 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
apnea hypopnea index after sildenafil vs. placebo | Hours

SECONDARY OUTCOMES:
Sleep parameters (latency, efficiency etc) following sildenafil vs. placebo | hours

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Ẕerifin, Israel